CLINICAL TRIAL: NCT03972215
Title: Effect of Berberine on Insulin Release at a High Blood Glucose Level in Normal Man
Brief Title: Berberine Hyperglycemic Clamp
Acronym: BBR HC
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Jin-Kui Yang (Other)
Responsible Party: Sponsor-Investigator, Jin-Kui Yang, Professor, PhD, Beijing Tongren Hospital
Organization: Beijing Tongren Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: BBR CLAMP
Record Dates: First submitted 2019-05-29; First posted 2019-06-03 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Diabetes Mellitus
Keywords: Hyperglycemic Clamp
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Berberine treatment (Experimental)
  Interventions: Drug: Berberine Chloride; Drug: Placebo
- Placebo control (Placebo Comparator)
  Interventions: Drug: Berberine Chloride; Drug: Placebo

INTERVENTIONS:
Drug: Berberine Chloride — Traditional Chinese Medicine
Drug: Placebo — Placebo Control

SUMMARY:
Berberine (BBR) is a traditional Chinese medicine used to treat diabetes mellitus for thousands of years in China. The glucose-lowering effect of BBR has been confirmed in numerous studies. Nevertheless, the detailed mechanisms of action through which BBR exerts its effects are not yet fully elucidated. In previous data, Jin-Kui Yang found that BBR could promote insulin secretion in mice and isolated islets. In this current study, investigators plan to examine the insulinotropic effect of BBR in human through hyperglycemic clamp method.

ELIGIBILITY:
Inclusion Criteria:

1. Adult healthy male, aged ≥18 and ≤45 years old.
2. Subject/ legal representative is able to understand and sign informed consent form.
3. Body mass index (BMI) 18-25 kg/m2.
4. Normal oral glucose tolerance test prior to study.
5. No family history of diabetes mellitus.
6. No medication treatment within 4 weeks prior to baseline visit and during the study.
7. Willing and able to comply with all study-related procedures, including not incorporating significant changes in diet.

Exclusion Criteria:

1. Infection with hepatitis (A, B, or C), HIV and syphilis.
2. History of allergic reaction to berberine or any component in the formulation of the study drugs.
3. Cumulative amount of blood loss (eg. blood donation) over 400mL within 3 months prior to baseline visit and during the study.
4. Alcohol drinking within 2 weeks prior to baseline visit and during the study.
5. Use of illegal drugs or positive in urine drugs screen.
6. Smoke during the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-02-17 (Actual)

PRIMARY OUTCOMES:
Differences of serum insulin levels between BBR and placebo treatment groups during the 2-hour hyperglycemic clamp study. | Single dosage for one experiment and crossover repeat once after 2 weeks washout period
  To compare the mean serum insulin levels in the two groups during hyperglycemic clamp study.
Differences of serum C-peptide levels between BBR and placebo treatment groups during the 2-hour hyperglycemic clamp study. | Single dosage for one experiment and crossover repeat once after 2 weeks washout period
  To compare the mean serum C-peptide levels in the two groups during hyperglycemic clamp study.

SECONDARY OUTCOMES:
Differences of glucose infusion rates between BBR and placebo treatment groups during the 2-hour hyperglycemic clamp study. | Single dosage for one experiment and crossover repeat once after 2 weeks washout period
  To compare the mean glucose infusion rates in the two groups during hyperglycemic clamp study.
Differences of blood glucose levels between BBR and placebo treatment groups during the 2-hour hyperglycemic clamp study. | Single dosage for one experiment and crossover repeat once after 2 weeks washout period
  To compare the mean blood glucose levels in the two groups during hyperglycemic clamp study.

OTHER OUTCOMES:
Heart rate and QT-interval duration using electrocardiogram before and after drug treatment. | Single dosage for one experiment and crossover repeat once after 2 weeks washout period
  Electrocardiogram will be performed in subjects before and after drug treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhao MM, Lu J, Li S, Wang H, Cao X, Li Q, Shi TT, Matsunaga K, Chen C, Huang H, Izumi T, Yang JK. Berberine is an insulin secretagogue targeting the KCNH6 potassium channel. Nat Commun. 2021 Sep 23;12(1):5616. doi: 10.1038/s41467-021-25952-2. PMID 34556670